CLINICAL TRIAL: NCT05601180
Title: Interventional, Prospective, National, Multicentre, Randomised, Open-label, Controlled Clinical Study Comparing Two Parallel Groups, One Control Arm (Standard Treatment) Versus Intervention Arm (Standard Treatment + Study Product) Evaluating the Efficacy of Respicure® 0.38% /0.38% (Resveratrol / Quercetin) Phytotherapy Product From BEKER® Laboratories as an add-on Treatment in the Management of Respiratory Conditions Including Asthma (Partially Controlled),Chronic Obstructive Pulmonary Disease "COPD" (Stage A, B, C and D) and Long Coronavirus Disease "COVID" in Algerian Adult Patients .
Brief Title: Evaluation of the Efficacy of Respicure® (Resveratrol / Quercetin) in the Management of Respiratory Conditions Including Asthma,COPD and Long COVID.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beker Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RESPIRE DZ
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Long COVID
Keywords: Phytotherapy; Inhalation; Complementary medicine
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Post-Acute COVID-19 Syndrome; Respiratory Aspiration | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stadard of care (Active Comparator): standard treatment that is prescribed by the treating physician.
  Interventions: Other: Standard of care
- Standard of care + Respicure® (Experimental): standard treatment that is prescribed by the treating physician in addition to Respicure®
  Interventions: Other: Respicure®

INTERVENTIONS:
Other: Respicure® — Respicure® is an inhalation solution that contains two natural extracts: quercetin and resveratrol in a concentration of 0.38%/0.38%.
  Arms: Standard of care + Respicure®
Other: Standard of care — standard treatment is prescribed by the treating physician.
  Arms: Stadard of care

SUMMARY:
Interventional, Prospective, National, Multicentre, Randomised, Open-label, Controlled Clinical Study Comparing Two Parallel Groups, One Control Arm (Standard Treatment) Versus Intervention Arm (Standard Treatment + Study Product) Evaluating the Efficacy of Respicure® 0.38% /0.38% (Resveratrol / Quercetin) Phytotherapy Product From BEKER Laboratories as an add-on Treatment in the Management of Respiratory Conditions Including Asthma (Partially Controlled),COPD (Stage A, B, C and D) and long COVID in Algerian Adult Patients .

DETAILED DESCRIPTION:
This is an interventional, prospective, national, multicenteric, randomized, open-label, controlled clinical study comparing two arms: Control arm taking the standard of care Versus Intervention arm (standard of care + Respicure®).

A total of 480 patients (160 in each group of pathology i.e Asthme, COPD and long COVID, distributed through 8 centers resulting in 20 patients/center for each group of pathology). The administration of the study product is by randomaisation.The data will be collected during 5 visits for the two arms as following:

* Visit V1 on D0: inclusion, signature of informed consent and implementation of the RESPIRE DZ protocol with delivery to patients of a one-month supply of Respicure® for the intervention arm,
* Intermediary visit on D15: face-to-face and/or by telephone to assess safety after the use of Respicure® for the intervention arm.
* Visit V2 on D30: follow-up visit with delivery to patients of a one-month supply of Respicure® for the intervention arm,
* Visit V3 on D60: follow-up visit with delivery to patients of a one-month supply of Respicure® for the intervention arm,
* Visit V4 at D90:follow-up visit at the end of the use of the study product,
* Visit V5 at D180: follow-up and end-of-study visit.

ELIGIBILITY:
* Inclusion Criteria for Asthma patients:

  1. Male, female, aged ≥19.
  2. Being able to provide written informed consent before the study.
  3. Patient with partially controlled asthma: Assessment of asthma control over the month preceding the use of Respicure ® by a symptomatic assessment (Tick one or two symptoms):

  3. 1 Daytime symptoms more than twice a week, 3. 2 One or more nocturnal awakenings, 3. 3 Need for rescue medication more than twice a week, 3. 4 One or more activity limitations

  4. Patient followed for at least a year and mastering the technique of using devices i.e. aerosols, nebulizer etc…
* Inclusion Criteria for COPD patients:

  1. Male, female, ≥40 years old
  2. Being able to provide written informed consent before the study.
  3. Patient with COPD stage A, B, C or D in stable condition with no exacerbations in the past 4 weeks.
  4. Patient followed for at least a year and mastering the technique of using devices i.e. aerosols, nebulizer etc…
* Inclusion Criteria for long covid patients:

  1. Male, female, aged ≥19.
  2. Being able to provide written informed consent before the study.
  3. Patients followed for respiratory symptoms linked to long Covid (symptoms for more than 12 weeks).

Exclusion Criteria :

1. Patient with severe asthma (for asthma groupe only)
2. Prior use of Respicure®.
3. Concomitant use with the following products: cytochrome P450 3A4 substrate drugs (e.g. statin, antifungals and fexofenadine), antibiotics (quinolones), immunosuppressants (cyclosporine) and glycoprotein P substrate drugs, e.g. antifungal and antiarrhythmic .
4. Hypersensitivity to any of the ingredients.
5. Hypersensitivity to peanuts.
6. Concomitant intake of a product containing one or both of the active ingredients (resveratrol/quercetine).
7. Pregnancy/ lactation.
8. People who need to undergo surgery.
9. Participation in another clinical study within the previous 30 days.
10. Patient with asthma-COPD overlap syndrome or any other respiratory disease such as pneumonia, tuberculosis, pulmonary embolism, etc.
11. Hormone-sensitive conditions such as breast cancer, uterine cancer, ovarian cancer, endometriosis or uterine fibroids.
12. Patients requiring admission to intensive care and/or requiring respiratory assistance.
13. Patients requiring anticoagulant treatment at curative doses.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change of asthma symptoms in partially controlled patients . | Change from Baseline at 3 months
  The assessment of asthma management will be based on:
  1. Improvement in symptoms measured at baseline and during the follow-up period and results will be compared to those of the control group to determine asthma control using the following criteria:
  * Daytime symptoms at most twice a week,
  * No nocturnal awakenings,
  * Need for rescue medication at most twice a week,
  * No limitation of activities.
Change of COPD symptoms in patients with stage A, B, C or D. | Change from Baseline at 3 months
  The assessment of reduction in symptoms will be be compared to those of the control group and will be based on reducing CAT scoring "COPD assessment test" to be less than 10.
Change of COPD symptoms in patients with stage A, B, C or D. | Change from Baseline at 3 months.
  The assessment of reduction in symptoms will be based on reducing mMRC scoring "modified Medical Research Council" where 0 being the best and 4 being the worst.
Change of respiratory symptoms related to long COVID. | Change from Baseline at 3 months
  The assessment of the respiratory symptoms linked to long COVID will be based on the reduction in dyspnea and cough by measuring m mMRC scoring "modified Medical Research Council" where 0 being the best and 4 being the worst.
Change of respiratory symptoms related to long COVID. | Change from Baseline at 3 months
  The assessment of the respiratory symptoms linked to long COVID will be based on:
  - Improvement of Blood oxygen saturation.

SECONDARY OUTCOMES:
Tolerance | 3 months
  Tolerance to Respicure®: assessment of the occurrence of serious/non-serious adverse events during the study period.
Morbidity for Asthma patients | 3 months
  Minimisation or absence of hospitalisation and Reduction of number of exacerbations
Change of CAT scoring for Asthma patients | Change from Baseline at 3 months
  Improvement of CAT scoring (Asthma control test) more than 20.
Change of Respiratory function for Asthma patients | Change from Baseline at 3 months
  Evaluation of respiratory function by spirometry to detect Variation of PEF (Peak expiratory flow) compared to baseline (in %)
Change of Respiratory function for Asthma patients | Change from Baseline at 3 months
  Evaluation of respiratory function by spirometry to detect:
  Improved FEV1/FVC ratio (Forced expiratory volume in one second/ Forced vital capacity) compared to baseline (in %)
Change of Respiratory function for Asthma patients | Change from Baseline at 3 months
  Evaluation of respiratory function by spirometry to detect a decreased FEV1 (Forced expiratory volume in one second) variability compared to baseline (in %)
Morbidity & Exacerbations for COPD patients | 6 months
  Minimisation or absence of hospitalisation and The prevention of future exacerbations "time to onset of the 1st exacerbation in six (06) months",
Exacerbations for COPD patients | 6 months.
  The prevention of future exacerbations "time to onset of the 1st exacerbation in six (06) months",
Change of Respiratory function for COPD patients | Change from Baseline at 3 months
  Evaluation of respiratory function by spirometry to detect variation of PEF (Peak expiratory flow) compared to baseline (in %)
Change of Respiratory function for COPD patients | Change from Baseline at 3 months
  Evaluation of respiratory function by spirometry to detect variation of FEV (Forced expiratory volume) compared to baseline (in %)
Morbidity for long COVID patients | 6 months.
  Minimisation or absence of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Pr Mersak GHARNAOUT, Professor, Principal Investigator — CHU Beni Messous/ Pneumologie A
Locations (8):
- Algeria (8):
  - CHU Beni Messous/Pneumologie A, Algiers
  - CHU Beni Messous/Pneumologie B, Algiers
  - CHU Annaba/Pneumo-phtisiologie, Annaba
  - EPH Batna/Pneumo-phtisiologie, Batna City
  - CHU Constantine/Pneumo-phtisiologie, Constantine
  - EPH Laghouat/Pneumo-phtisiologie, Laghouat
  - CHU Oran/Pneumo-phtisiologie B, Oran
  - CHU Sidi Bel Abbes/Pneumo-phtisiologie, Sidi Bel Abbes

IPD SHARING:
Plan to Share IPD: No